CLINICAL TRIAL: NCT06985095
Title: Effectiveness of a Structured Nutrition Educational Program on Glycemic Control, Quality of Life, and Cardiovascular Risk in Patients With Uncontrolled Diabetes Using Multiple Daily Insulin Injections
Brief Title: Evaluation of a Structured Nutrition Educational Program in Insulin-treated Diabetic Patients in Vietnam
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cho Ray Hospital (Other)
Responsible Party: Principal Investigator, Ly Na Dau, Endocrinologist, Cho Ray Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChorayMUIN2025
Record Dates: First submitted 2025-05-05; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus
Keywords: nutrition educational program; diabetes; multiple daily injection insulin users
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (No Intervention): Participants in this arm only receive a nutrition booklet, written and designed by researchers. They don't join the lessons with the researcher.
- Nutrition Intervention group (Experimental): Intervention group receives the same booklet and attends four monthly lessons with a researcher about healthy eating for diabetes.
  Interventions: Other: Nutrition educational program

INTERVENTIONS:
Other: Nutrition educational program — Participants in the intervention group will attend a structured nutrition education program consisting of four monthly sessions, each lasting approximately 40 to 60 minutes. These sessions will be conducted in small groups by the researcher.
  Each session includes: A 20-30 minute presentation delivered by the researcher using visual aids, such as slides and educational images. A 20-30 minute interactive discussion to address participants' questions, clarify concepts.
  Session Topics:
  Treatment Goals in Diabetes Care: Overview of blood glucose targets and the importance of achieving glycemic control.
  Key Nutritional Components of Food: Roles of carbohydrates, proteins, fats, fiber, and their impact on blood glucose.
  Principles of Meal Planning: Adjusting energy intake based on physical activity levels and BMI.
  Understanding the Food Exchange System: Introduction to food exchange lists; selecting the appropriate number of food exchanges to meet individual energy needs.
  Arms: Nutrition Intervention group

SUMMARY:
The purpose of this study is to find out if learning about healthy eating can help people with diabetes control their blood sugar better.

This study is for men and women between 18 and 70 years old who use insulin at least twice a day but still have high blood sugar.

We want to answer the following questions:

Can nutrition education help lower HbA1c (a blood test that shows average blood sugar over the past 3 months)? Can it improve knowledge about nutrition, quality of life, and make blood sugar more stable? Will it help reduce fasting blood sugar, lipid levels, body weight, and the number of times low blood sugar (hypoglycemia) happens?

Participants will be divided into two groups:

One group will receive a nutrition booklet. The other group will receive the same booklet and join four monthly lessons with a researcher.

The four lessons will talk about:

Goals for managing diabetes Main nutrients in food How to plan meals How to eat in a way that supports better blood sugar control

DETAILED DESCRIPTION:
This study will involve 115 people with diabetes who need to take insulin at least twice a day. It includes those who already use multiple insulin injections but still have high blood sugar, and those who are newly switched to at least two insulin shots daily because their blood sugar is not well controlled with pills or pills plus one injection.

The study will take place at Cho Ray Hospital in Ho Chi Minh City, Vietnam, and will run from 2025 to the end of 2026. People will be invited to join at the Endocrinology Consultation Unit. If they agree, their phone number will be collected and the research team will call them later to explain more about the study. If they are still interested, they'll be asked to keep a food diary for three days before their screening.

On the screening day, they'll sign a short consent form, get blood tests to check their sugar, HbA1c, cholesterol, and kidney function, talk with a nutrition researcher about their food diary, and have a usual consultation with their doctor. If they meet all the criteria and agree to take part, they'll sign the full consent form and take short tests on nutrition knowledge and quality of life. The quality of life questionnaire used is the SF-36 questionnaire, and nutrition knowledge is assessed using the Diabetes-related Nutrition Knowledge Questionnaire (DRNK-Q).

After that, they will be randomly assigned to one of two groups. One group will get a nutrition booklet only. The other group will receive the booklet plus attend four monthly sessions with a researcher to learn about healthy eating for diabetes. In each group, 10 participants will also wear a flash glucose monitor (a small device that checks sugar levels without finger pricks) three times: at the beginning, after 3 months, and after 6 months. These participants will be selected based on age, HbA1c level, ability to use the device, and whether they often experience low blood sugar.

During the 6-month study period, all participants will have blood tests every 3 months to check HbA1c, fasting sugar, and lipid; they will be asked monthly about any low blood sugar episodes; they will repeat the nutrition and quality of life tests at 6 months; their weight and waist size will be measured every 3 months, and their height will be measured at the start of the study

ELIGIBILITY:
Inclusion Criteria:

* People between 18 and 70 years old.
* People who come to Cho Ray Hospital for diabetes care and plan to keep getting care there for at least six months.
* People who have diabetes and have been prescribed diabetes medicine.
* People who were recently diagnosed with diabetes, based on the latest guidelines from the American Diabetes Association.
* People whose blood sugar (HbA1c) level is higher than 8%.
* People who are currently using at least two insulin injections a day or have just started a daily multiple insulin injection plan because their diabetes is not well controlled.

Exclusion Criteria:

* People who are seriously ill and need to stay in the hospital, such as those with infections, pneumonia, heart attacks, strokes, or infected diabetic foot.
* People who have cancer, serious mental health problems, or problems with drug use.
* People who do not want to take part or cannot follow the study plan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
the difference in the change of HbA1c between the two groups after six months of follow-up | For enrollment to the end of study at 6 months
  We will check each person's HbA1c level before starting the program, and then again every three months. After six months, we will look at how much each person's HbA1c has changed compared to the beginning. Then we'll compare the average change between the two groups using a statistical test.

SECONDARY OUTCOMES:
The changes in quality of life after six months of follow-up within and between groups | From enrollment to the end of study at 6 months
  Quality of life will be assessed at the start of the study and again after six months using the SF-36 questionnaire. The total scores from the questionnaire will be calculated, and the average change in scores will be compared between the two groups.
The change in nutrition knowlege at the start of the study and after 6 months between two groups | From enrollment to the end of study at 6 months.
  Nutrition knowledge will be assessed using the Diabetes-related Nutrition Knowledge questionnaire (DRNK-Q) at the start of the study and again after six months. The mean change in total score of the questionnaire before and after six months will be compared between the two groups. The maximum score is 27 for the people who consume alcohol, and is 25 for the people who don't consume alcohol. The minimum score is zero. The higher score indicates an improvement in nutritional knowledge.
The changes in BMI (Body mass index) after six months of follow-up within and between groups | From enrollment to the end of treatment at 6 months
  BMI will be measured at the beginning of the study and every three months. Changes in this health indicator over time will be tracked within each group, and the average changes over six months will be compared between the two groups.
The changes in Waist Circumference after six months of follow-up within and between groups | From enrollment to the end of treatment at 6 months
  Waist Circumference will be measured at the beginning of the study and every three months. Changes in this health indicator over time will be tracked within each group, and the average changes over six months will be compared between the two groups.
The changes in plasma LDL cholesterol (bad cholesterol) after six months of follow-up within and between groups | From enrollment to the end of treatment at 6 months
  Plasma LDL cholesterol (bad cholesterol) will be measured at the beginning of the study and every three months. Changes in this health indicator over time will be tracked within each group, and the average changes over six months will be compared between the two groups.
The changes in plasma total cholesterol after six months of follow-up within and between groups | From enrollment to the end of treatment at 6 months
  Plasma total cholesterol will be measured at the beginning of the study and every three months. Changes in this health indicator over time will be tracked within each group, and the average changes over six months will be compared between the two groups.
The changes in plasma triglycerides after six months of follow-up within and between groups | From enrollment to the end of treatment at 6 months
  Plasma triglycerides will be measured at the beginning of the study and every three months. Changes in this health indicator over time will be tracked within each group, and the average changes over six months will be compared between the two groups.
The changes in plasma HDL cholesterol (good cholesterol) after six months of follow-up within and between groups | From enrollment to the end of treatment at 6 months
  Plasma HDL cholesterol (good cholesterol) will be measured at the beginning of the study and every three months. Changes in these health indicators over time will be tracked within each group, and the average changes over six months will be compared between the two groups.

OTHER OUTCOMES:
The change in total daily insulin dose before and after the intervention between groups | From enrollment to the end of study at six months
  The total daily insulin dose will be collected each month. The changes in total daily insulin before and six months after the intervention of the two groups will be compared.
The change in time in range over six months between groups: standard group and nutrition intervention group | From enrollment to the end of study at six months
  We assess blood glucose fluctuations using a flash continuous glucose monitoring system at the start of the study and then every three months for six months. The mean change in time in range within groups will be assessed and compared across the groups.
The change in the number of insulin injections per day before and after the intervention between groups | From enrollment to the end of treatment at 6 months
  The number of insulin injections per day will be collected each month. The changes in the number of insulin injections per day before and six months after the intervention of the two groups will be compared.
The change in the number of anti-diabetic oral medications before and after the intervention between groups | From enrollment to the end of treatment at 6 months
  the number of anti-diabetic oral medications will be collected each month. The change in the number of anti-diabetic oral medications before and six months after the intervention of the two groups will be compared
The change in time in hyperglycemia over six months between groups: standard group and nutrition intervention group | From enrollment to the end of treatment at 6 months
  The mean change in time in hyperglycemia in each group will be assessed and compared between groups.
The change in time in hypoglycemia over six months between groups: standard group and nutrition intervention group | From enrollment to the end of treatment at 6 months
  The mean change in time in hypoglycemia each groups will be assessed and compared across groups.

CONTACTS AND LOCATIONS:
Overall Officials: Na Ly Dau, MD, Principal Investigator — Cho Ray Hospital
Locations (1):
- Cho Ray Hospital, Ho Chi Minh City, Vietnam, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data (IPD) collected during the study will be made publicly available upon reasonable request or through a designated open-access repository after publication of the main results. Data will be shared in compliance with ethical approvals and participant consent, ensuring that no personally identifiable information is disclosed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available during

REFERENCES:
- [Background] Bowen ME, Cavanaugh KL, Wolff K, Davis D, Gregory RP, Shintani A, Eden S, Wallston K, Elasy T, Rothman RL. The diabetes nutrition education study randomized controlled trial: A comparative effectiveness study of approaches to nutrition in diabetes self-management education. Patient Educ Couns. 2016 Aug;99(8):1368-76. doi: 10.1016/j.pec.2016.03.017. Epub 2016 Mar 19. PMID 27026388
- [Background] Speight J, Amiel SA, Bradley C, Heller S, Oliver L, Roberts S, Rogers H, Taylor C, Thompson G. Long-term biomedical and psychosocial outcomes following DAFNE (Dose Adjustment For Normal Eating) structured education to promote intensive insulin therapy in adults with sub-optimally controlled Type 1 diabetes. Diabetes Res Clin Pract. 2010 Jul;89(1):22-9. doi: 10.1016/j.diabres.2010.03.017. Epub 2010 Apr 18. PMID 20399523
- [Background] Trento M, Trinetta A, Kucich C, Grassi G, Passera P, Gennari S, Paganin V, Tedesco S, Charrier L, Cavallo F, Porta M. Carbohydrate counting improves coping ability and metabolic control in patients with Type 1 diabetes managed by Group Care. J Endocrinol Invest. 2011 Feb;34(2):101-5. doi: 10.1007/BF03347038. Epub 2010 May 3. PMID 20440106
- [Background] Schmidt S, Schelde B, Norgaard K. Effects of advanced carbohydrate counting in patients with type 1 diabetes: a systematic review. Diabet Med. 2014 Aug;31(8):886-96. doi: 10.1111/dme.12446. PMID 24654856
- [Background] Franz MJ, MacLeod J, Evert A, Brown C, Gradwell E, Handu D, Reppert A, Robinson M. Academy of Nutrition and Dietetics Nutrition Practice Guideline for Type 1 and Type 2 Diabetes in Adults: Systematic Review of Evidence for Medical Nutrition Therapy Effectiveness and Recommendations for Integration into the Nutrition Care Process. J Acad Nutr Diet. 2017 Oct;117(10):1659-1679. doi: 10.1016/j.jand.2017.03.022. Epub 2017 May 19. No abstract available. PMID 28533169
- [Background] Franz MJ, Monk A, Barry B, McClain K, Weaver T, Cooper N, Upham P, Bergenstal R, Mazze RS. Effectiveness of medical nutrition therapy provided by dietitians in the management of non-insulin-dependent diabetes mellitus: a randomized, controlled clinical trial. J Am Diet Assoc. 1995 Sep;95(9):1009-17. doi: 10.1016/S0002-8223(95)00276-6. PMID 7657902
- [Background] Coppell KJ, Kataoka M, Williams SM, Chisholm AW, Vorgers SM, Mann JI. Nutritional intervention in patients with type 2 diabetes who are hyperglycaemic despite optimised drug treatment--Lifestyle Over and Above Drugs in Diabetes (LOADD) study: randomised controlled trial. BMJ. 2010 Jul 20;341:c3337. doi: 10.1136/bmj.c3337. PMID 20647285
- [Background] Kitajima Y, Mikami N, Hyodo T, Hida M, Kawakami J. Carbohydrate Counting: A Simple Method of Dietary Management for Glycemic Control in Japanese Diabetic Hemodialysis Patients. Contrib Nephrol. 2017;189:262-269. doi: 10.1159/000451045. Epub 2016 Dec 12. PMID 27951578
- [Background] Laurenzi A, Bolla AM, Panigoni G, Doria V, Uccellatore A, Peretti E, Saibene A, Galimberti G, Bosi E, Scavini M. Effects of carbohydrate counting on glucose control and quality of life over 24 weeks in adult patients with type 1 diabetes on continuous subcutaneous insulin infusion: a randomized, prospective clinical trial (GIOCAR). Diabetes Care. 2011 Apr;34(4):823-7. doi: 10.2337/dc10-1490. Epub 2011 Mar 4. PMID 21378215
- [Background] Cadario F, Prodam F, Pasqualicchio S, Bellone S, Bonsignori I, Demarchi I, Monzani A, Bona G. Lipid profile and nutritional intake in children and adolescents with Type 1 diabetes improve after a structured dietician training to a Mediterranean-style diet. J Endocrinol Invest. 2012 Feb;35(2):160-8. doi: 10.3275/7755. Epub 2011 May 27. PMID 21623150
- [Background] Powers MA, Gal RL, Connor CG, Mangan M, Maahs DM, Clements MA, Mayer-Davis EJ. Eating patterns and food intake of persons with type 1 diabetes within the T1D exchange. Diabetes Res Clin Pract. 2018 Jul;141:217-228. doi: 10.1016/j.diabres.2018.05.011. Epub 2018 May 26. PMID 29772288
- [Background] DAFNE Study Group. Training in flexible, intensive insulin management to enable dietary freedom in people with type 1 diabetes: dose adjustment for normal eating (DAFNE) randomised controlled trial. BMJ. 2002 Oct 5;325(7367):746. doi: 10.1136/bmj.325.7367.746. PMID 12364302
- [Background] Andrews RC, Cooper AR, Montgomery AA, Norcross AJ, Peters TJ, Sharp DJ, Jackson N, Fitzsimons K, Bright J, Coulman K, England CY, Gorton J, McLenaghan A, Paxton E, Polet A, Thompson C, Dayan CM. Diet or diet plus physical activity versus usual care in patients with newly diagnosed type 2 diabetes: the Early ACTID randomised controlled trial. Lancet. 2011 Jul 9;378(9786):129-39. doi: 10.1016/S0140-6736(11)60442-X. Epub 2011 Jun 24. PMID 21705068
- [Background] Franz MJ, Powers MA, Leontos C, Holzmeister LA, Kulkarni K, Monk A, Wedel N, Gradwell E. The evidence for medical nutrition therapy for type 1 and type 2 diabetes in adults. J Am Diet Assoc. 2010 Dec;110(12):1852-89. doi: 10.1016/j.jada.2010.09.014. PMID 21111095
- [Background] Holt RIG, DeVries JH, Hess-Fischl A, Hirsch IB, Kirkman MS, Klupa T, Ludwig B, Norgaard K, Pettus J, Renard E, Skyler JS, Snoek FJ, Weinstock RS, Peters AL. The management of type 1 diabetes in adults. A consensus report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetologia. 2021 Dec;64(12):2609-2652. doi: 10.1007/s00125-021-05568-3. PMID 34590174